CLINICAL TRIAL: NCT05924256
Title: A Phase II Study of Advanced Salivary Gland Carcinoma Based on Molecular Typing
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associate Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGC-IIT-umbrella
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Salivary Gland Carcinoma
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): This arm for HER2-positive salivray gland carcinoma.
  Interventions: Drug: SHR-A1811
- Arm 2 (Experimental): This arm for AR-postive salivray gland carcinoma.
  Interventions: Drug: SHR 3680 + leuprolide
- Arm 3： 3a adenoid cystic carcinoma and 3b non-adenoid cystic carcinoma (Experimental): This arm for salivray gland carcinoma without HER-2 alteration or AR-postive.
  Interventions: Drug: SHR-A1921
- Arm 4 (Experimental): This arm for low HER2 expression salivray gland carcinoma.
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811
  Arms: Arm 1
Drug: SHR 3680 + leuprolide — SHR 3680 + leuprolide
  Arms: Arm 2
Drug: SHR-A1921 — SHR-A1921
  Arms: Arm 3： 3a adenoid cystic carcinoma and 3b non-adenoid cystic carcinoma
Drug: SHR-A1811 — SHR-A1811
  Arms: Arm 4

SUMMARY:
This is a single-center, open-label, phase 2 study to evaluate the efficacy and safety of target therapy for patients with relapsed/metastastic salivary gland carcinoma based on molecular typing.

DETAILED DESCRIPTION:
Patients with IHC HER2 IHC 3+ or IHC 2+/ISH+ will be located into arm 1 to receive anti-her2 ADC（SHR- A1811） Patients with IHC AR positive will be located into arm 2 to receive anti-androgen therapy (SHR-3680)+leuprolide Patients with HER2 negative and AR negative will be located into arm 3 to receive anti-TROP2 ADC (SHR-A1921) Patients with IHC HER2 IHC 1+ or IHC 2+/ISH- will be located into arm 4 to receive anti-her2 ADC（SHR- A1811）

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. Aged ≥ 18 but ≤ 75 years, male or female;
3. Histologically confirmed to be locally advanced or metastatic salivary gland carcinoma;
4. Arm1: salivary gland carcinoma patients with HER-2 overexpression ； Arm 2: salivary gland carcinoma patients with AR-positive; Arm 3: salivary gland carcinoma patients without HER-2 alteration or AR-positive; Arm 4: salivary gland carcinoma patients with low HER-2 expression;
5. At least one measurable lesion (according to RECIST v1.1, long diameter of measurable lesion scanned by spiral CT should be ≥ 10 mm or short diameter of swollen lymph node should be ≥ 15 mm; according to RECIST vl.1 standards, a previously treated lesion with local treatment can be used as target lesions after clear progress);
6. ECOG Perfomance Status: 0~1;
7. Estimated survival time ≥ 12 weeks;
8. The main organs function are normal, and meet the following requirements (within 7 days before the start of study treatment):

   Blood routine examination(no blood transfusion within 14 days before screening, no granulocyte colony stimulating factor (G-CSF), no medication corrected):1) Hemoglobin (HB)≥ 90g / L;2) Neutrophil count (ANC) ≥ 1.5 × 109 / L;3) platelets (PLT) ≥ 80 × 109 / L; Blood biochemical tests are subject to the following criteria (no albumin is delivered 14 days prior to screening):1) Serum total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); 2) alanine aminotransferase (ALT), aspartate aminotransferase (AST])< 2.5 × ULN; if liver metastasis, ALT and AST ≤ 5 × ULN;3) Serum creatinine (Cr) ≤ 1 × ULN or endogenous creatinine clearance > 50ml / min (Cockcroft-Gault formula); International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeds the range of normal controls ≤ 6 seconds; Urine protein <2+ (if urine protein ≥ 2+, 24-hour urine protein can be quantified, 24-hour urine protein quantitation <1.0g can be included);
9. Women of childbearing age must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and volunteer to use appropriate methods during the observation period and within 8 weeks after the last study drug administration; for men, sterilization surgery should be performed, or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug;
10. Patient who are expected to have good compliance and can accept follow-up visit for the efficacy and adverse reactions according to the program requirements.

Exclusion Criteria:

1. Have other active malignancies within 5 years or at the same time. Localized tumors that have been cured, such as cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ, can be enrolled.
2. Other anti-tumor treatments (including but not limited to chemotherapy, radiotherapy, etc.) were used within 28 days prior to the first use of the study drug. if the last dose of anti-tumor drug had been stopped ≥ 5 half-life can be allowed.
3. There are clinical symptoms or diseases of the heart that are not well controlled, such as:

   According to the New York Heart Association (NYHA) standard, level II or higher cardiac dysfunction or echocardiography: left ventricular ejection fraction<50%; unstable angina; Myocardial infarction occurred within 1 year before the start of treatment; Clinically significant supraventricular or ventricular arrhythmia that requires treatment or intervention; corrected QT interval(QTc) > 450ms (male); QTc > 470ms (female) (Calculation of QTc interval with Fridericia formula; if the QTc is abnormal, it can be detected three times at an interval of 2 minutes, and the average value is taken);
4. Patients with high blood pressure who cannot be reduced to normal range by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (average of BP based on ≥2 measurements), allowing the use of antihypertensive treatment to achieve the above parameters.
5. A variety of factors that affect the absorption of oral medications (such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction) (Only apply for Arm 2 patients);
6. Patients with a risk of gastrointestinal bleeding may not be enrolled, including the following: (1) active digestive ulcer lesions, and fecal occult blood (++); (2) those with a history of melena and hematemesis within 3 months;
7. Abnormal coagulation function (INR>1.5×ULN,activated partial thromboplastin time>1.5×ULN), with bleeding tendency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | at the end of every 2 cycles(for arm1, arm3 and arm4, each cycle is 21 days, for arm2, each cycle is 28 days)
  Objective response rate defined as the patients confirmed complete response or partial response under RECIST 1.0 criteria.

SECONDARY OUTCOMES:
DCR | at the end of every 2 cycles(for arm1, arm3 and arm4, each cycle is 21 days, for arm2, each cycle is 28 days)
  DCR defined as the patients confirmed complete response or partial response or stable disease under RECIST 1.0 criteria.
Progression-free Survival (PFS) | up to 2 years
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival (OS) | up to 2 years
  Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.
Adverse events | Since the signing of informed consent forms to 30 days after the last cycle
  Hematologic and non hematologic adverse event (CTCAE 5.0）

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, Doctor, Principal Investigator — Fudan University
Locations (1):
- Dongmei Ji, Shanghai, China

IPD SHARING:
Plan to Share IPD: No